CLINICAL TRIAL: NCT05554770
Title: Prevalence of Positional Nystagmus in a Population of Healthy Adults
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dan Dupont Hougaard, MD, Associate Professor, Aalborg University Hospital
Other Study IDs: N-20220034; F2022-081 (Registry Identifier: Datatilsynet, Region Nordjylland, Denmark)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Positional Nystagmus; Healthy Volunteers
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Examinations in a TRV chair — Positional tests (Dix-Hallpike and SRT) traditionally used to diagnose BPPV uwith a TRV chair.

SUMMARY:
To investigate the prevalence of positional nystagmus in a population of healthy Danish adults.

DETAILED DESCRIPTION:
Open-label, cross-sectional prospective study examining the prevalence of positional nystagmus in healthy adults (adult with no previous or current inner ear disease) using a mechanical repositioning chair (TRV-chair, Interacoustics, Middelfart, Denmark). Patients will undergo traditional testing related to positional nystagmus by means of both the Dix-Hallpike test and Supine Roll Test (SRT) bilaterally. Latency, duration, and slow phase velocities will be registered and examiner as well as order of the positional tests performed with the TRV chair will be block randomized.

ELIGIBILITY:
Inclusion Criteria:

* + 18 years

Exclusion Criteria:

* Previous or current BPPV, inner ear disease, other ear conditions or neurological conditions
* Reduced eye mobility
* Alcohol consumption within 48 hours
* Weight > 150 kg.
* Known cerebral aneurysm
* Cerebral haemorrhage within 1 month
* Trouble cooperating during examinations
* DHI-score > 14

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A population of healthy adults who meets the in- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of positional nystagmus | 2 years
  Number of subjects presenting with positional nystagmus during specific changes of head positions.

SECONDARY OUTCOMES:
Characteristics of positional nystagmus | 2 years
  Description the characteristics (latency, velocity, duration, direction) of positional nystagmus in healthy subjects.

OTHER OUTCOMES:
Specify current diagnostic criteria for Benign Paroxysmal Positional Vertigo | 2 years
  Expansion and clarification of current diagnostic criteria for BPPV

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Hougaard, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Otolaryngology, Head- and Neck Surgery and Audiology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No